CLINICAL TRIAL: NCT01072305
Title: Einfluss Der Intermittierenden Pneumatischen Kompression Der Unteren Extremitäten Auf Den Intraoperativen Flüssigkeitsbedarf
Brief Title: Pneumatic Compression of the Legs to Reduce Fluid Demand in Minor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: Masimo Corp. (loan of medical devices) (Unknown); Villa Sana GmbH (loan of medical devices) (Unknown)
Responsible Party: Prof. Dr. med. Andreas Hoeft, Dept. of Anesthesiology and Intensive care, medical center of the Rheinische-Friedrich-Wilhelms-Universität Bonn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAIIPC01
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-01

CONDITIONS: ENT Surgery
Keywords: fluid restriction; fluid therapy; intraoperative care
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent pneumatic compression (IPC) (Experimental): IPC from induction of general anesthesia to completion of skin closure.
  Interventions: Device: Intermittent pneumatic compression (IPC)
- control (Placebo Comparator): IPC - placebo from induction of general anesthesia to closure of the skin
  Interventions: Device: IPC - placebo

INTERVENTIONS:
Device: Intermittent pneumatic compression (IPC) — Intermittent pneumatic compression (sequential compression) using a cuff consisting of 12 chambers inflated sequentially from forefoot to groin with decremental inflation pressures (60-38 mmHg), pressure release after complete inflation, and reinflation after 4 seconds pause. ICP cuffs are covered with a frame and drapes for blinding purpose.
  Other Names: Lympha Press plus (Model 1033 EL), SN 0248; Cuffs: adult
  Arms: Intermittent pneumatic compression (IPC)
Device: IPC - placebo — ICP cuffs are placed next to/between legs and covered with a frame and drapes for blinding purpose. IPC device is run fom induction of general anesthesia to closure of the skin.
  Other Names: Lympha Press plus (Model 1033 EL), SN 0248; Cuffs: adult
  Arms: control

SUMMARY:
Fluid restriction has become of great interest in perioperative care. There is, however, a conflict of interest between fluid restriction and hemodynamic stability. The investigators hypothesized that intermittent pneumatic compression may recruit blood from venous capacity vessels of the lower limbs and thus enable fluid restriction without compromising hemodynamic stability.

DETAILED DESCRIPTION:
Induction of general anesthesia has a variety of effects on the cardiovascular system, all resulting in impaired hemodynamics. Besides reduced sympathetic tone (Sellgren et al.;Ebert, Kanitz, and Kampine) and direct negative inotropic effect of anesthetic agents(Gare et al.), reduction of cardiac preload (Dahlgren et al.;von Spiegel et al.) plays a major role. Therefore administration of large amounts of i.v. fluid is a common method to counter adverse hemodynamic effects. In addition, substitution for fluid loss during preoperative fasting has been recommended for decades. However, preoperative fasting may lead to less fluid loss than assumed so far(Jacob et al.), and there is increasing evidence that i.v. fluid has many adverse effects. Perioperative weight gain due to fluid overload is an independent predictor of mortality (Lowell et al.). Besides a detrimental effect on gastrointestinal (Nisanevich et al.;Gan et al.;Noblett et al.;Wakeling et al.;Lobo et al.), i.v. fluid may harm the endothelial barrier (Bruegger et al.), possibly leading to a vicious circle of impaired barrier function and increased demand for i.v. fluids (Chappell et al.).

In order to restore cardiac preload, timing, volume, and composition of the fluid are important. Free water (e.g. glucose 5%) or "physiologic saline" have very high volumes of distribution, while colloid application is associated with various adverse effects (Schramko et al.;Dart et al.). This has led to increased interest in intraoperative volume restriction (de Aguilar-Nascimento et al.;McArdle et al.;Muller et al.;Walsh et al.). The ideal i.v. fluid remains to be found, yet it exists already if autotransfusion is considered as fluid therapy. The recruitable amount of blood that is contained in capacity vessels of the legs has not been precisely determined, but estimates range from 100 to 300 ml in each leg (citations). The easiest way to recover the blood that is sequestered from systemic circulation is passive leg raising or Trendelenburg positioning, two methods that have entered intensive care routine to assess volume responsiveness. However in many clinical situations passive leg raising or Trendelenburg position is not feasible, e.g. ear, nose, and throat (ENT) or neurosurgical procedures. Intermittent pneumatic compression (IPC) is an established therapeutic intervention for several indications such as lymphedema, post thrombotic ulcers and arterial claudication (Wienert et al.)and has been recommended for intraoperative prevention of thrombembolism. (Geerts et al.). When used during laparoscopy it can effectively reduce hemodynamic adverse effects of pneumoperitoneum (Alishahi et al.;Bickel et al.;Bickel et al.;Bickel et al.;Kurukahvecioglu et al.). So far its use in a general surgical population to promote volume restriction has not been assessed. We compared fluid demand in patients undergoing minor ENT surgery with or without IPC under a standardized, goal-directed fluid management protocol.

ELIGIBILITY:
Inclusion Criteria:

* minor ENT surgery without anticipated relevant blood loss

Exclusion Criteria:

* ASA Status > II
* contraindication to IPC
* unwillingness or inability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Intraoperative fluid demand | intraoperative
  Intraoperative = from induction of general anesthesia to end of the surgical procedure, length of procedure may vary (expected mean duration= 45 min)

SECONDARY OUTCOMES:
hemodynamic stability | intraoperative
local complications of compression therapy | perioperative
  perioperative = from induction of general anesthesia (= beginning of compression therapy) to discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hoeft, Professor, Principal Investigator — Department of Anesthsiology and Intensive Care, Medical Centerof the Rheinische Friedrich-Wilhelms-University of Bonn
Locations (1):
- Medical center of the Rheinische Friedrich Willhelm Univesity of Bonn, Bonn, Germany